CLINICAL TRIAL: NCT00438516
Title: Follow-up of Families in Early Preventive Intervention
Acronym: MemphisYear9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: David Olds, Principal Investigator, University of Colorado Denver
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01HD043492 (NIH); 5R01MH061428-02 (NIH)
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2007-12

CONDITIONS: Child Rearing; Adolescent Development; Reproductive Behavior; Risk Reduction Behavior
Keywords: home visits; pregnancy; welfare; child development; mortality
MeSH Terms: conditions — Reproductive Behavior; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control group
- 2 (Experimental): Nurse home visitation
  Interventions: Behavioral: nurse home visitation

INTERVENTIONS:
Behavioral: nurse home visitation — Nurse home visits from midway through pregnancy to child age 2
  Arms: 2

SUMMARY:
This project supports the post-third-grade assessment of 693 children and their families who were enrolled in a randomized trial of a program of prenatal and infancy home visitation by nurses that was epidemiologically and theoretically grounded. The project will determine whether the beneficial effects of the program on maternal, child, and family functioning extend through the early elementary school years, giving particular attention to maternal life-course and children's emerging antisocial behavior. Assessments of the children will be based on both mother and teacher reports. Teachers are independent, natural raters of the children's adaptation to an important social context. There are numerous reasons to expect that, from a developmental perspective, the effects of the program will increase as children experience the increased academic demands associated with entry into third grade. In addressing these questions, the current study will determine the extent to which this program of prenatal and infancy home visitation by nurses can produce enduring effects on maternal and child functioning (giving particular attention to the prevention of early-onset disruptive behavior disorders) in urban African Americans that are consistent with those achieved with whites in a central New York state county in a separate trial of this program conducted over the past 20 years.

DETAILED DESCRIPTION:
This project supports the post-third-grade assessment of 693 children and their families who were enrolled in a randomized trial of a program of prenatal and infancy home visitation by nurses that was epidemiologically and theoretically grounded. The sample enrolled was composed of low-income women who had no previous live births and who were largely African American (92%), unmarried (98%), and adolescent (67%) at the time of registration during pregnancy. In earlier phases of assessment, the program was found to improve the quality of care patients provided to their children, to reduce children's health-care encounters in which injuries were detected, to increase children's sequential processing skills as measured by the KABC, to reduce the number of dysregulated aggressive and violent themes expressed in their response to the MacArthur Story Stem Battery, and so to improve maternal life-course as reflected in fewer subsequent pregnancies, reduced use of welfare, and increases in the marriage and cohabitation with the biological father of the child. Many of the benefits in the area of parental care-giving and child functioning were concentrated in those children and their mothers who had few psychological resources (where psychological resources was defined as the absence of mental disorder symptoms, adequate intellectual functioning, and belief in their control over their life circumstances).

The project will determine whether the beneficial effects of the program on maternal, child, and family functioning extend through the early elementary school years, giving particular attention to maternal life-course and children's emerging antisocial behavior. Assessments of the children will be based on both mother and teacher reports. Teachers are independent, natural raters of the children's adaptation to an important social context. There are numerous reasons to expect that, from a developmental perspective, the effects of the program will increase as children experience the increased academic demands associated with entry into third grade. In addressing these questions, the current study will determine the extent to which this program of prenatal and infancy home visitation by nurses can produce enduring effects on maternal and child functioning (giving particular attention to the prevention of early-onset disruptive behavior disorders) in urban African Americans that are consistent with those achieved with whites in a central New York state county in a separate trial of this program conducted over the past 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Women <29 weeks of gestation were recruited if they had no previous live births, no specific chronic illnesses thought to contribute to fetal growth retardation or pre-term delivery, and at least 2 of the following socio-demographic risk conditions:

  * Unmarried,
  * <12 years of education, and
  * Unemployed.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2000-06; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
interval between birth of first and second children; | When first child was 9
cumulative subsequent births per year following birth of the first child through the first child's 9th birthday; | When first child was 9
duration of mother's relationship with current partner; | When first child was 9
being partnered with, cohabiting with, or married to the child's biological father; | When first child was 9
her sense of mastery; | When first child was 9
duration of use of welfare (AFDC and TANF) and food stamps per year following birth of the first child; | When first child was 9
the counts of maternal arrests and days jailed, | When first child was 9
the count of substances used (3 or more drinks of alcohol 3 or more times per month in the last year, use of marijuana, and use of cocaine since last interview at child age 6) | When first child was 9
children's grade point averages in reading, math, and behavior (conduct) from their school records | At child age 9
children's achievement test scores | At child age 9
teacher report of antisocial behavior | At child age 9
maternal report of child disruptive behavior disorders and depressive and anxiety disorders | At child age 9

SECONDARY OUTCOMES:
counts of subsequent miscarriages, abortions, and low-birth-weight newborns; | When first child was 9
women's reported participation in the workforce; | When first child was 9
their depression; | When first child was 9
whether they had experienced physical violence from any of their partners since their first child was 6; | When first child was 9
and the portion of time their current partners were employed while they were together following birth of the first child | When first child was 9
number of times children were retained in grades 1-3 | At child age 9
placement in special education | At child age 9
teachers' assessments of children's behavior | At child age 9
children's deaths | By child age 9

CONTACTS AND LOCATIONS:
Overall Officials: David L Olds, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Rochester School of Nursing, Rochester, New York, United States

REFERENCES:
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Kitzman H, Olds DL, Sidora K, Henderson CR Jr, Hanks C, Cole R, Luckey DW, Bondy J, Cole K, Glazner J. Enduring effects of nurse home visitation on maternal life course: a 3-year follow-up of a randomized trial. JAMA. 2000 Apr 19;283(15):1983-9. doi: 10.1001/jama.283.15.1983. PMID 10789666
- [Background] Kitzman H, Olds DL, Henderson CR Jr, Hanks C, Cole R, Tatelbaum R, McConnochie KM, Sidora K, Luckey DW, Shaver D, Engelhardt K, James D, Barnard K. Effect of prenatal and infancy home visitation by nurses on pregnancy outcomes, childhood injuries, and repeated childbearing. A randomized controlled trial. JAMA. 1997 Aug 27;278(8):644-52. PMID 9272896
- [Result] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740